#### **Trial Protocol**

A multi-centre randomized, placebo-controlled trial of mirabegron, a new beta3-adrenergic receptor agonist on the progression of left ventricular mass and diastolic function in patients with structural heart disease

# BETA3\_LVH

Coordinating investigator

Prof. Jean-Luc Balligand

Full professor, Head of Department

Pharmacology and Therapeutics (FATH)

Avenue Mounier, 52, B1.53.09

1200 Brussels, Belgium

Phone: +32-2-7645260/+32-2-7645262

Fax: +32-2-7645269

Biometry

Dr. Oana Brosteanu, Dr. Dirk Hasenclever

Clinical Trial Centre Leipzig

Universität Leipzig Härtelstraße 16-18.

04107 Leipzig, Germany

Phone: +49-341-97 16 250

Fax: +49-341-97 16 189

Sponsor

UNIVERSITÉ CATHOLIQUE DE LOUVAIN
PLACE DE L'UNIVERSITE 1, 1348 LOUVAIN LA NEUVE, Belgium

Date: November 3<sup>rd</sup>, 2016

Version: Final 5.0

EudraCT-Nr.: 2015-003146-75

Clinical Trials.gov identifier: NCT02599480

ISRCTN-Number: ISRCTN65055502

© Version 08 valid as of 01 January 2013

Print: [xxx]

Written by/authors:

Based on the protocol template from the Zentrum für Klinische Studien Leipzig - KKS.

## **Table of Contents**

| | | PAGE |
|---|---|---|
| GENE | RAL INFORMATION | 6 |
| | onsible Parties | |
| Synop | sislule of Assessments and Procedures | 10 |
| 1 | RATIONALE | |
| 1.1<br>1.2<br>1.3 | Medical BackgroundRationaleRisk-Benefit Considerations | |
| 2 | OBJECTIVES | ERREUR! SIGNET NON DEFINI. |
| 2.1<br>2.2 | Primary ObjectiveSecondary Objectives | |
| 3 | TRIAL DESIGN AND DESCRIPTION | ERREUR! SIGNET NON DEFINI. |
| 3.1<br>3.2 | Trial DesignRequirements at the Trial Sites regarding Pe non défini. | rsonnel and Equipment <b>Erreur! Signet</b> |
| 3.3<br>3.4<br>3.5 | Trial Sites and Number of Trial Subjects Expected Duration of Trial Premature Termination of the Trial | |
| 4 | TRIAL SUBJECTS | ERREUR! SIGNET NON DEFINI. |
| 4.1<br>4.2<br>4.3<br>4.4<br>4.5<br>4.6 | Inclusion Criteria | ppulations ividuals |
| 5 | INVESTIGATIONAL PRODUCT | ERREUR ! SIGNET NON DEFINI. |
| 5.1<br>5.2<br>5.3<br>5.4<br>5.5 | Trial DrugsPackaging and Labelling of the Trial Drug Drug AccountabilityAdministration of the Study DrugBlinding and Unblinding | <br><br> |
| 6 | INDIVIDUAL TRIAL PROCEDURES | ERREUR ! SIGNET NON DEFINI. |
| 6.1<br>6.2<br>6.3<br>6.4 | Patient Information and Informed Consent Enrolment in the Trial Description of the Treatment Procedures Premature Termination of the Therapy for Inc. défini. | <br> |
| 6.5<br>6.6 | Premature study termination for individual pa Plan for Further Treatment | |
| 7 | METHODS OF DIAGNOSTICS AND DATA S<br>DEFINI. | SAMPLINGERREUR! SIGNET NON |
| 8 | ADVERSE EVENTS (AE/SAE) | ERREUR ! SIGNET NON DEFINI. |
| ឧ 1 | Adverse Events (AF) | Erreur I Signet non défini |

| | Cofety Analysis | Frank I Cianat non défini |
|---|---|---|
| 8.2<br>8.3 | Safety Analysis Concomitant Diseases | |
| 8.4 | Serious Adverse Events (SAE) | |
| 8.5 | Periodic Reports | |
| 8.6 | Suspected Unexpected Serious Adverse Reactions (St | |
| 8.7 | Other Safety Relevant Issues | |
| 8.8 | Therapeutic Procedures | |
| 8.9 | Dealing with Pregnancy | |
| 9 | BIOMETRY ERR | |
| 9.1 | Biometrical Aspects of the Trial Design | |
| 9.2 | End Points | |
| 9.3<br>9.4 | Statistical Description of the trial hypothesis | |
| 9. <del>4</del><br>9.5 | Statistical Methods | |
| 9.6 | Statistical Monitoring | |
| 9.7 | Interim Analysis | • |
| 9.8 | Final Analysis | |
| 10 | CONCOMITANT SCIENTIFIC PROJECTS ERR | <del>-</del> |
| 10.1 | Endothelial Function/Pulse amplitude tonometry and m Signet non défini. | easurement of HbNO Erreur! |
| 10.2 | Abundance/activity of brown/beige fat | |
| 10.3 | Analysis of blood and urine samples for scientific purpo | ses related to cardiac disease |
| 11 | ETHICAL, LEGAL AND ADMINISTRATIVE ASPECTS DEFINI. | SERREUR! SIGNET NON |
| 11.1 | GCP-Statement | Erreur ! Sianet non défini. |
| 11.1<br>11.2 | GCP-StatementInitial Submission | |
| 11.2 | Initial Submission Protocol AmendmentsERR | <br><br>REUR! SIGNET NON DEFINI. |
| 11.2<br>11.3 | Initial Submission Protocol AmendmentsERR | <br><br>REUR! SIGNET NON DEFINI. |
| 11.2<br>11.3<br><b>12</b><br>12.1<br>12.2 | Initial Submission Protocol Amendments DOCUMENTATION ERR Case Report Forms (CRF) Data Management | <br><br>REUR! SIGNET NON DEFINI.<br><br> |
| 11.2<br>11.3<br><b>12</b><br>12.1 | Initial Submission Protocol Amendments DOCUMENTATION ERR Case Report Forms (CRF) | <br><br>REUR! SIGNET NON DEFINI.<br><br> |
| 11.2<br>11.3<br><b>12</b><br>12.1<br>12.2 | Initial Submission. Protocol Amendments DOCUMENTATION ERR Case Report Forms (CRF) Data Management Archiving. SUPERVISION OF THE CLINICAL TRIAL ERR | REUR! SIGNET NON DEFINI REUR! SIGNET NON DEFINI. |
| 11.2<br>11.3<br><b>12</b><br>12.1<br>12.2<br>12.3<br><b>13</b> | Initial Submission Protocol Amendments DOCUMENTATION | REUR! SIGNET NON DEFINI REUR! SIGNET NON DEFINI |
| 11.2<br>11.3<br><b>12</b><br>12.1<br>12.2<br>12.3<br><b>13</b><br>13.1<br>13.2 | Initial Submission Protocol Amendments DOCUMENTATION | REUR! SIGNET NON DEFINI REUR! SIGNET NON DEFINI |
| 11.2<br>11.3<br><b>12</b><br>12.1<br>12.2<br>12.3<br><b>13</b><br>13.1<br>13.2<br>13.3 | Initial Submission. Protocol Amendments DOCUMENTATION | REUR! SIGNET NON DEFINI REUR! SIGNET NON DEFINI. REUR! SIGNET NON DEFINI |
| 11.2<br>11.3<br><b>12</b><br>12.1<br>12.2<br>12.3<br><b>13</b><br>13.1<br>13.2<br>13.3<br>13.4 | Initial Submission. Protocol Amendments DOCUMENTATION | REUR! SIGNET NON DEFINI REUR! SIGNET NON DEFINI. REUR! SIGNET NON DEFINI |
| 11.2<br>11.3<br><b>12</b><br>12.1<br>12.2<br>12.3<br><b>13</b><br>13.1<br>13.2<br>13.3<br>13.4<br>13.5 | Initial Submission Protocol Amendments DOCUMENTATION ERR Case Report Forms (CRF) Data Management Archiving. SUPERVISION OF THE CLINICAL TRIAL ERR Access to Source Data Monitoring Audits Inspections Independent Supervision of the Trial | EUR! SIGNET NON DEFINI. EUR! SIGNET NON DEFINI. |
| 11.2<br>11.3<br><b>12</b><br>12.1<br>12.2<br>12.3<br><b>13</b><br>13.1<br>13.2<br>13.3<br>13.4 | Initial Submission. Protocol Amendments DOCUMENTATION | EUR! SIGNET NON DEFINI. EUR! SIGNET NON DEFINI. |
| 11.2<br>11.3<br><b>12</b><br>12.1<br>12.2<br>12.3<br><b>13</b><br>13.1<br>13.2<br>13.3<br>13.4<br>13.5 | Initial Submission. Protocol Amendments DOCUMENTATION | EUR! SIGNET NON DEFINI. EUR! SIGNET NON DEFINI. |
| 11.2<br>11.3<br><b>12</b><br>12.1<br>12.2<br>12.3<br><b>13</b><br>13.1<br>13.2<br>13.3<br>13.4<br>13.5<br><b>14</b> | Initial Submission Protocol Amendments DOCUMENTATION ERR Case Report Forms (CRF) Data Management Archiving. SUPERVISION OF THE CLINICAL TRIAL ERR Access to Source Data Monitoring. Audits Inspections Independent Supervision of the Trial DATA PROTECTION AND CONFIDENTIALITY ERR Declaration regarding Data Protection Declaration regarding the Pseudonymized Transfer of Inon défini. | EUR! SIGNET NON DEFINI. EUR! SIGNET NON DEFINI. |
| 11.2<br>11.3<br><b>12</b><br>12.1<br>12.2<br>12.3<br><b>13</b><br>13.1<br>13.2<br>13.3<br>13.4<br>13.5<br><b>14</b> | Initial Submission. Protocol Amendments DOCUMENTATION | EUR! SIGNET NON DEFINI. EUR! SIGNET NON DEFINI. |
| 11.2<br>11.3<br>12<br>12.1<br>12.2<br>12.3<br>13.1<br>13.2<br>13.3<br>13.4<br>13.5<br>14.1<br>14.2 | Initial Submission Protocol Amendments DOCUMENTATION Case Report Forms (CRF) Data Management Archiving SUPERVISION OF THE CLINICAL TRIAL Access to Source Data Monitoring Audits Inspections Independent Supervision of the Trial DATA PROTECTION AND CONFIDENTIALITY Declaration regarding Data Protection Declaration regarding the Pseudonymized Transfer of Inon défini. ADMINISTRATIVE AGREEMENTS ERR Adherence to the Protocol | EUR! SIGNET NON DEFINI. EUR! SIGNET NON DEFINI. EUR! SIGNET NON DEFINI. |
| 11.2<br>11.3<br><b>12</b><br>12.1<br>12.2<br>12.3<br><b>13</b><br>13.1<br>13.2<br>13.3<br>13.4<br>13.5<br><b>14</b><br>14.1<br>14.2<br><b>15</b><br>15.1<br>15.2 | Initial Submission Protocol Amendments DOCUMENTATION ERR Case Report Forms (CRF) Data Management Archiving. SUPERVISION OF THE CLINICAL TRIAL Access to Source Data Monitoring. Audits Inspections Independent Supervision of the Trial DATA PROTECTION AND CONFIDENTIALITY. ERR Declaration regarding Data Protection Declaration regarding the Pseudonymized Transfer of Inon défini. ADMINISTRATIVE AGREEMENTS ERR Adherence to the Protocol Funding and Insurance | EUR! SIGNET NON DEFINI. EUR! SIGNET NON DEFINI. EUR! SIGNET NON DEFINI. |
| 11.2<br>11.3<br>12<br>12.1<br>12.2<br>12.3<br>13.1<br>13.2<br>13.3<br>13.4<br>13.5<br>14.1<br>14.2 | Initial Submission Protocol Amendments DOCUMENTATION Case Report Forms (CRF) Data Management Archiving SUPERVISION OF THE CLINICAL TRIAL Access to Source Data Monitoring Audits Inspections Independent Supervision of the Trial DATA PROTECTION AND CONFIDENTIALITY Declaration regarding Data Protection Declaration regarding the Pseudonymized Transfer of Inon défini. ADMINISTRATIVE AGREEMENTS ERR Adherence to the Protocol | EUR! SIGNET NON DEFINI. EUR! SIGNET NON DEFINI. EUR! SIGNET NON DEFINI. |

| 16 | REFERENCES | ERREUR ! SIGNET NON DEFINI. |
|---|---|---|
| 17 | PROTOCOL SIGNATURES | ERREUR ! SIGNET NON DEFINI. |
| 18 | PROTOCOL AGREEMENT | ERREUR ! SIGNET NON DEFINI. |
| 19 | APPENDIX | ERREUR ! SIGNET NON DEFINI. |
| 19.1<br>19.2<br>19.3<br>19.4 | DefinitionsAcronyms | |
| List | of Tables | |
| table 1 | 1: Schedule of Assessments and Procedu | res |
| List | of Figures | |
| Figure | 1: Flowchart of the trial | |
| Figure | 2: Sample of blister-label | |
| Figure | 3. Sample of box-label | Frreur ! Signet non défini |

## **GENERAL INFORMATION**

#### **Responsible Parties**

| Sponsor (according to Belgian drug law) | Université catholique de Louvain (UCL) Place de l'Université 1 1348 Louvain la Neuve Belgium Authorised representative of the sponsor, Promotor: Prof. Jean-Luc Balligand |
|---|---|
| Coordinating investigator(s) | Prof. Dr. Jean-Luc Balligand Full professor, Head of Department Pharmacology and Therapeutics (FATH) Avenue Mounier, 52, B1.53.09 1200 Brussels, Belgium Phone: +32-2-7645260/+32-2-7645262 Fax: +32-2-7645269 E-Mail: jean-luc.balligand@uclouvain.be |
| Deputy of Coordinating investigator | Anne-Catherine Pouleur Cliniques universitaires Saint-Luc Avenue Hippocrate, 10 1200 Bruxelles, Belgique Phone: +32-2-764 28 12, Fax: +32-2-764 89 80 E-Mail: anne-catherine.pouleur@uclouvain.be |
| Project Management | Dr Ir Nancy van Overstraeten UCL-FATH Institut de Recherche Expérimentale et Clinique (IREC) Building Vésale 5th floor ; 52 Avenue Mounier B1.53.09; 1200 Brussels; Belgium Phone: +32-2-764 52 88 Fax: +32-2-764 5269 E-Mail: nancy.vanoverstraeten@uclouvain.be Dr. Petra Neuhaus Zentrum für Klinische Studien Leipzig – KKS Universität Leipzig Härtelstraße 16-18, 04107 Leipzig, Germany Phone: +49 341 97 16255 Fax: +49 341 97 16 16189 E-Mail: petra.neuhaus@zks.uni-leipzig.de |
| Pharmacovigilance | Madlen Dörschmann<br>Zentrum für Klinische Studien Leipzig – KKS<br>Universität Leipzig |

| | Härtelstraße 16-18, 04107 Leipzig, Germany<br>Phone: +49 341 97 16129<br>Fax: +49 341 97 16 16278<br>E-Mail: madlen.doerschmann@zks.uni-leipzig.de |
|---|---|
| Data Management | Angelika Beyer Zentrum für Klinische Studien Leipzig – KKS Universität Leipzig Härtelstraße 16-18, 04107 Leipzig, Germany Phone: +49 341 97 16261 Fax: +49 341 97 16259 E-Mail: angelika.beyer@zks.uni-leipzig.de |
| Biometry | Dr. Oana Brosteanu Zentrum für Klinische Studien Leipzig – KKS Universität Leipzig Härtelstraße 16-18, 04107 Leipzig, Germany Phone: +49 341 97 16251 Fax: +49 341 97 16189 E-Mail: oana.brosteanu@zks.uni-leipzig.de Dr. Dirk Hasenclever Institut für Medizinische Informatik, Statistik und Epidemiologie Universität Leipzig Härtelstraße 16-18, 04107 Leipzig, Germany Phone: +49 341 97 16121 Fax: +49 341 97 16109 E-Mail: dirk.hasenclever@imise.uni-leipzig.de |
| Monitoring | Nicole Köppe-Bauernfeind Zentrum für Klinische Studien Leipzig – KKS Universität Leipzig Härtelstraße 16-18, 04107 Leipzig, Germany Phone: +49 341 97 16266 Fax: +49 341 97 16259 E-Mail: nicole.koeppe-bauernfeind@zks.uni-leipzig.de |
| Funding | EU Framework Programme for Research and Innovation, Horizon 2020: Mr. Grzegorz OWSIANIK Marie-Christine Groenen Medical research and the challenge of ageing European Commission DIRECTORATE-GENERAL FOR RESEARCH & INNOVATION Medical research and the challenge of ageing Directorate Health |

| | B-1049 Brussels Belgium |
|---|---|
| | Phone: +32 22951192 E-Mail: Grzegorz.OWSIANIK@ec.europa.eu Marie-Christine.Groenen@ec.europa.eu |
| | Organisation: Prof. Dr. Stefan Anker Charité - Universitätsmedizin Berlin Campus Virchow-Klinikum Augustenburger Platz 1, 13353 Berlin, Germany Phone: +49 (0) 30-450 553463 Fax: +49 (0) 30-450 553951 E-Mail: s.anker@cachexia.de |
| | Chair: Karl Swedberg, Prof. MD Department of Molecular and Clinical Medicine, Sahlgrenska Academy, University of Gothenburg, Sweden, and National Heart and Lung Institute, Imperial College, London, UK E-mail: karl.swedberg@gu.se |
| Data Safety and Monitoring Board | Members: Dan Atar, MD, FESC, FACC, FAHA Professor of Cardiology Head of Research, Div. of Medicine Oslo University Hospital, Ullevål Kirkeveien 166, Building 3-A N - 0407 Oslo - Norway Ph: + 47 22 11 91 00 Email W: dan.atar@ous-hf.no Email H: dan.atar@online.no |
| | Luigi Tavazzi, MD, FESC, FACC GVM Care and Research, E.S. Health Science Foundation, Maria Cecilia Hospital Via Corriera, 1 48010 Cotignola (RA) - Emilia-Romagna Italy E-mail: 'Elisa Ghizzardi GVM Care&Research' <direzionescientifica-mch@gvmnet.it></direzionescientifica-mch@gvmnet.it> |
| | Hans Wedel KB Biostatistics Apelsingatan 115 |

| | 426 54 Västra Frölunda<br>Phone: 070-829 72 88<br>E-mail : hans.wedel@biostat.se |
|---|---|
| Concomitant scientific projects | Endothelial Function/Pulse amplitude tonometry and measurement of HbNO: Dr Ignatios Ikonomidis,MD,PhD,FESC Assistant Professor, Member of EACVI Nucleus member of ESC WG Peripheral Circulation 2nd Cardiology Department University of Athens Attikon Hospital Rimini 1, 12462 Haidari, Greece E-mail: ignoik@otenet.gr,ignoik@gmail.com tel +30 6944805732 fax +30 210 5832351 ,210 5832192 Abundance/activity of brown/beige fat: Dr Renaud Lhommel (CUSL) Cliniques universitaires Saint-Luc Avenue Hippocrate, 55 bte B1.55.01 1200 Bruxelles Belgique Phone: +32 2 764 25 82 Fax: +32 2 764 16 02 E-Mail: renaud.lhommel@uclouvain.be |

# Synopsis

| Title of the trial | A multi-centre randomized, placebo-controlled trial of mirabegron, a new beta3-adrenergic receptor agonist on the progression of left ventricular mass and diastolic function in patients with structural heart disease. |
|---|---|
| Acronym | BETA3_LVH |
| Indication | Structural heart disease at high risk for progressive hypertrophic cardiac remodeling at risk of developing HFpEF (heart failure with preserved ejection fraction). |
| | The primary objective is to evaluate the effect of mirabegron (a new $\beta$ 3-specific agonist) on change in left ventricular mass and/or changes in diastolic function after 12 months of treatment in patients with cardiac structural remodeling with or without symptoms of heart failure (maximum NYHA II). |
| Primary goal of the trial / primary end point | <ul> <li>Two equally ranked, primary endpoints: <ul> <li>Change in left ventricular mass index (LVMI in g/m², defined as left ventricular mass divided by body surface) measured at baseline and 12 months after randomisation.</li> </ul> </li> <li>Change in diastolic function, assessed as the ratio of peak early transmitral ventricular filling velocity to early diastolic tissue Doppler velocity (E/e²) measured at baseline and 12 months after randomisation.</li> </ul> |
| | Effect of mirabegron on other indicators for diastolic heart disease, i.e. cardiac fibrosis, left atrial volume index, diastolic function (E/e'), maximal exercise capacity and laboratory markers (analysed after 6 or 12 months of mirabegron treatment). |
| Secondary goals of the trial / secondary end points | <ul> <li>Secondary endpoints: <ul> <li>Further MRI endpoints (all measured in the central MRI core lab)</li> <li>Cardiac fibrosis at baseline and at 12 months. Fibrosis is a key pathogenic mechanism of diastolic dysfunction, which is at the origin of HFpEF</li> <li>Left atrial volume index at baseline and at 12 months. This parameter determines diastolic filling (and was shown to predict treatment efficacy in HFpEF in the J-DHF trial (Yamamoto et al. 2013))</li> <li>LV mass index (by cardiac MRI) at 6 months,</li> <li>Diastolic function (E/e') at 6 months;</li> </ul> </li> <li>Laboratory parameters at baseline and at 3, 6 and 12 months <ul> <li>serum biomarkers (Galectin3, GDF15, NT-proBNP, hsTnT)</li> <li>metabolic parameters (fasting glucose, modified HOMA test, HbA1c, serum lipids)</li> </ul> </li> <li>Maximal exercise capacity (peak VO2) at baselineand 12 months.</li> </ul> |

| | Safety endpoints Incidence, severity and frequency of adverse and serious adverse events Mortality |
|---|---|
| Trial design | Two armed, prospective, randomized, placebo-controlled, multi-centric international phase IIb trial |
| | <ul> <li>Inclusion criteria: <ul> <li>Age between 18 and 90 years</li> <li>Morphological signs of structural cardiac remodelling by echocardiography, i.e. increased LV mass index (≥95 g/m² or higher for female; ≥115 g/m² or higher for male subjects (Ponikowski et al. 2016)) or end-diastolic wall thickness ≥13 mm in at least one wall segment</li> <li>Written informed consent</li></ul></li></ul> |
| Trial population | <ul> <li>Major exclusion criteria:</li> <li>Unstable arterial hypertension with systolic BP≥160 mm Hg and/or diastolic BP≥100 mm Hg (confirmed at three consecutive office measurements in sitting position); if so, the patient may be re-screened after optimization of anti-hypertensive treatment</li> <li>Hypertensive patients not under stable therapy according to current guideline algorithm (Mancia et al. 2013) (including stable medication for at least 4 weeks before inclusion)</li> <li>Documented ischemic cardiac disease: <ul> <li>current angina pectoris or</li> <li>ischemia on stress test or</li> <li>untreated coronary stenosis &gt;50% or</li> <li>history of acute myocardial infarction (AMI) or</li> <li>coronary artery bypass graft (CABG, &lt; than 3 months prior to screening) or</li> <li>percutaneous transluminal coronary angioplasty (PTCA) less than 3 months prior to screening.</li> </ul> </li> <li>Patients with uncontrolled recurrent persistent and permanent atrial fibrillation (AF) according to AHA/ACC/ESC guidelines (Dixon et al. 2005) (with a heart rate &gt; 100/min, RACE II - (Groenveld et al. 2013, 2013)). If AF with HR&gt;100/min, the patient may be rescreened after treatment for rate control.</li> <li>History of hospitalization for overt heart failure within last 12 months</li> <li>History of high degree impulse conduction blocks (&gt; 2nd degree AV block type 2)</li> <li>Patients after heart transplantation</li> <li>Genetic hypertrophic or dilated cardiomyopathy</li> <li>Dysthyroidism</li> </ul> |

- Severe valvulopathy (less than 1 cm2 aortic valve area, mitral insufficiency of severe grade at Doppler echo)
- · Congenital valvulopathies
- Patients with a known history of QT prolongation (QT>450ms) or patients with documented QT prolongation (QT>450 ms) while taking medicinal products known to prolong the QT interval.
- NYHA-class > II
- BMI >  $40 \text{ kg/m}^2$
- EF < 50%, regardless of symptoms
- Known other cause (i.e. COPD) of respiratory dysfunction; patients under positive pressure (CPAP) treatment for sleep apnea syndrome may be included, provided they have been efficiently controlled by CPAP for at least one year before inclusion in the study
- Moderate renal impairment defined as eGFR < 30 ml/min</li>
- Abnormal liver function tests (AST or ALT >2 X upper normal limit or patients with known hepatic impairment defined as Child-Pugh class B or higher)
- Type I diabetes, complicated type II diabetes (i.e. with documented coronary macroangiopathy, cfr exclusion criterion 1 or documented other vascular complication) (National Diabetes Education Initiative - NDEI).
- Patients with anemia (male: Hb <130 g/l, female: Hb <120 g/l)</li>
- · Patients with bladder outlet obstruction
- Patients using antimuscarinic cholinergic drugs for treatment of OAB
- Current use of digitalis, bupranolol, propranolol, nebivolol (known to interfere with β3AR signalling)
- Note: patients are allowed to take a β(1-2)-blocker, other than the drugs listed above (for explanation, see chapter ).
- Patients continuously treated with Sildenafil or other PDE5 inhibitors.
- Current use of antifungal azole derivatives (fluconazole, itraconazole, miconazole, posaconazole, voriconazole) (known inhibitors of CYP3A4, the main metabolizer of mirabegron)
- Current treatment with mirabegron or indication for future treatment with mirabegron due to other indications
- Contraindication for MRI (e.g.defibrillator, ferromagnetic devices or severe claustrophobia, pacemaker - the latter only, if MRI is contraindicated)
- · Pregnant or nursing women
- Women of child bearing potential without highly effective contraceptive measures (Clinical Trial Facilitation Group (CTFG) 9/15/2014):
  - combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
  - progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
  - intrauterine device (IUD)

| | <ul> <li>intrauterine hormone-releasing system ( IUS)</li> <li>bilateral tubal occlusion</li> <li>vasectomised partner</li> <li>sexual abstinence (only if in agreement with the preferred and usual lifestyle of the subject)</li> <li>while participating in the trial. There are no known interactions of the trial medication and hormone-based methods of contraception. In particular, no clinically relevant interactions have been observed when mirabegron was co-administered with therapeutic doses of a combined oral contraceptive medicinal product containing ethinylestradiol and levonorgestrel.</li> <li>Participation in any other interventional trial</li> <li>Patients unable to give informed consent (people under legal guardianship)</li> <li>Patients placed in an institution by official or court order</li> <li>Contraindication to mirabegron (e.g. hypersensitivity) or any other components of the trial medication</li> </ul> |
|---|---|
| Sample size | 296 patients overall (148 patients per treatment arm) will be randomised |
| Therapy | Experimental group: Administration of 50 mg mirabegron once daily per os (Betmiga®, Astellas Pharma) over a period of 12 months. Control group: Administration of placebo once daily per os over a period of 12 months. Verum and placebo will be manufactured by: Pharmacy of the University Hospital Leipzig Liebigstr. 20 D-04103 Leipzig |
| Biometry | Primary endpoints: Confirmatory analysis follows the intention to treat principle as close as possible and will be based on the full analysis set. In each patient, the primary endpoints will be assessed thrice: at the baseline visit, and at the 6 months and 12 months visits. Analyses of both primary endpoints are identically structured: Mean changes from baseline mean will be analysed using a repeated measurement linear mixed model without intercept containing the fixed, categorical effects of visit (baseline, 6 months, 12 months), treatment (verum / placebo), treatment by visit interaction Atrial fibrillation (yes / no), Diabetes mellitus (yes / no), as well as a patient-specific, visit random effect (3-dimensional normal with a general unstructured variance covariance matrix). |

| | Secondary endpoints: All other MRI and echocardiographic endpoints as well as peak VO2 will be analysed along the same lines as the primary endpoints. Time courses of metabolic parameters and specific biomarkers will be described. Adverse and serious adverse events will be compared by chi-square tests. Odds ratios with 95% confidence intervals will be provided. |
|---|---|
| | Individual treatment period: 12 months treatment per patient with an additional follow-up-phone visit at month 13 |
| Trial Duration | Trial: First patient in: April 2016 Patient-screening and recruitment: 33 months Last patient out (planned): December 2019 Final analysis (planned) December 2020 |